CLINICAL TRIAL: NCT06364995
Title: Effects of Specialised Physical Education in Volleyball on Middle School Students' Physical Fitness and Performance in Sichuan Province
Brief Title: Effects of Specialised Physical Education in Volleyball on Middle School Students' Physical Fitness and Performance
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Putra Malaysia (Other)
Responsible Party: Principal Investigator, MAO YIMOU, Principal Investigator, Universiti Putra Malaysia
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Basic Science
Other Study IDs: JKEUPM-2023-1364
Record Dates: First submitted 2024-03-31; First posted 2024-04-15 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Physical Fitness; Performance
Keywords: physical fitness; performance; Volleyball specialised physical education

STUDY DESIGN:
Intervention Model Description: In this experiment, the experimental group used the intervention of specialised physical education teaching of volleyball. However, the control group only conducted traditional physical education teaching content
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Volleyball specialised physical education (Experimental): Volleyball specialised physical education intervention in weeks 1-10 of the experiment
  Interventions: Behavioral: Volleyball
- Traditional Physical Education (Active Comparator): This arm is the control group receiving a traditional Physical Education program， Over 10 weeks, participants will engage in regular physical education sessions that include volleyball training
  Interventions: Behavioral: Traditional Physical Education

INTERVENTIONS:
Behavioral: Volleyball — Volleyball Specialised Physical Education Intervention is a step-by-step approach to teaching the intervention. Each lesson was conducted as a Warm-up (10 minutes), Basic contents of the PE lesson (25 minutes), and Cool-down (5 minutes). From the learning of basic skills in the first session to the final Combination Practice underhand service, receive, service, pass, spiking, and block, from the simple to the difficult, the intensity of the training is from weak to strong, Allowing participants to build upon a solid foundation toward mastering intricate volleyball maneuvers. Intensity modulation is key to this intervention; training intensity evolves from moderate to vigorous, aligning with the increasing complexity of skills and the physical demand required to execute them proficiently. The curriculum is thoughtfully designed to transition from basic skill execution to complex gameplay, with each lesson introducing new skills or refining existing ones.
  Arms: Volleyball specialised physical education
Behavioral: Traditional Physical Education — Participants participating in the control group will attend traditional physical education classes following the established physical education syllabus. Participants in the control group will attend four 40-minute classes per week over ten weeks. Each session will consist of a warm-up (10 minutes), the basics of PE (25 minutes), and a cool-down (5 minutes). The duration and intensity of the experimental and control groups were the same, which allowed for a better comparison.
  Arms: Traditional Physical Education

SUMMARY:
Physical education stands as a collaborative, bilateral activity essential for the development and improvement of young people's physical qualities and plays a pivotal role in youth sports promotion. Volleyball offers a blend of aerobic and anaerobic exercises, developing muscle strength, bone density, cardiovascular health, and fine-tuning the nervous system. It is effective in improving physical attributes such as strength, speed, agility, endurance, and coordination, which are crucial for holistic student development and success in the standardized PE entrance examinations for senior high school.

Recent trends have highlighted a decline in physical fitness among youth, as evidenced by rising obesity rates and increasing failure rates in fitness assessments. To counteract this, the Ministry of Education of the People's Republic of China 2021 has initiated a shift towards "specialised physical education," integrating health knowledge with basic and specialised motor skills training. This innovative educational model hopes to improve student physical fitness across educational tiers.

Therefore, this study chose volleyball specialised physical education as an intervention to study the effect of physical fitness and The PE entrance examination for senior high school performance of middle school students.

DETAILED DESCRIPTION:
This study employed a Cluster Randomized Controlled Trial (CRCT) design, conducted across two middle schools in Chengdu City, Sichuan Province, China. The investigators systematically assigned an experimental group to undergo a meticulously structured 10-week specialised volleyball physical education program, tailored according to rigorous research protocol. Parallel to this, the control group participated in a traditional physical education curriculum.

The experimental group engaged in a targeted training regimen focused on elevating volleyball competencies. The program was carefully segmented into four distinct developmental phases, ensuring a gradual and measurable enhancement of skills. Each session maintained strict adherence to a prescribed intensity gradient, incorporating exercises that evolved from low to high intensity, simple to complex executions, and individual techniques to holistic gameplay.

The intervention unfolded as follows:

Warm-up (10 min): A series of dynamic activities designed to prepare the body for rigorous physical activity, emphasizing mobility and injury prevention.

Basic contents of PE lesson (25 min): This segment included a progressive suite of volleyball drills and exercises, fine-tuned to fortify foundational skills during the initial weeks and gradually introducing strategic elements as the weeks advanced. Skill refinement, tactical understanding, and technical proficiency were paramount throughout the phases.

Cool-down (5 min): Post-training activities focused on lowering heart rate and stretching to aid recovery, reduce muscle soreness, and improve flexibility.

The four progressive phases of the intervention were as follows:

Phase 1 (1-2 weeks) Foundational Technique Acquisition Phase 2 (3-5 weeks) Skill Refinement and Expansion Phase 3 (6-8 weeks) Advanced Techniques and Tactical Application Phase 4 (9-10 weeks) Competitive Play and Specialisation.

To measure the impact of this intervention, pre-test was conducted to establish baseline data before the experiment, and post-test was delivered after the tenth week. The testing protocol aimed to capture the progression in both physical fitness and proformance, providing a comparative analysis between the specialised physical education intervention and traditional physical education approach.

ELIGIBILITY:
Inclusion Criteria:

1. Age and Education Level: Must be third-year students currently enrolled in a junior middle school.
2. Need Students who took The PE entrance examination forsenior high school performance in Sichuan Province.
3. Health Status: confirming the absence of any acute illnesses or physical impairments that could impair test performance.
4. Physical Ability: Must be capable of performing all test activities designed for the study.

Exclusion Criteria:

* 1. Chronic Organ Diseases: Students with a documented history of chronic organ diseases, such as liver cirrhosis, chronic kidney disease, or others that could impact physical performance or require ongoing medical intervention, are excluded.

  2. Cardiovascular Conditions: Students with any form of heart disease, including but not limited to congenital heart defects, arrhythmias, or history of myocardial infarction, are excluded.

  3. Chronic Illness: Students with any chronic illnesses that could impair their ability to participate fully in the physical tests or that could be exacerbated by physical exertion, including but not limited to asthma, severe allergies, or diabetes requiring insulin management, are excluded.

  4. Physical Disabilities: Students with congenital disabilities or physical impairments that prevent full participation in the study's required physical activities are excluded. This includes, but is not limited to, mobility impairments, significant musculoskeletal disorders, or other conditions that limit physical activity or exercise capacity.

  5. Medical: Students must not have any medical conditions or take any medications that, in the opinion of a medical professional, would make participation in the study unsafe or interfere with the interpretation of the test results.

Ages: 13 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 90 (Estimated)
Dates: Start 2024-01-10 (Actual); Primary Completion 2024-06-28 (Estimated); Study Completion 2024-07-05 (Estimated)

PRIMARY OUTCOMES:
Effects of physical fitness of middle school students | Pretest: Before experiment;Post test:10 weeks end
  By the physical fitness ,all the test outcomes and testing content are assessed using the "National Physical Fitness Test Standards for Students" China, 2014. The tests included are Spirometry Testing (FVC), 800m Run for Girls / 1000m Run for Boys, 1-minute Sit-Ups for Girls / Pull-Ups for Boys, Standing Long Jump Test, and Body Mass Index (BMI). Participants undergo an initial test before the intervention begins, and a retest after the 10-week intervention period. The researcher will conduct these tests according to assessment metrics, all test results are standardized quantification according to the "National Physical Fitness Test Standards for Students" China, 2014,and the test results are classified into four levels: 10-50 points (fail), 60-78 points (pass), 80-85 points (good), and 90-100 points (excellent).
Effects on middle school students' PE entrance examination for senior high school test performance | Pretest: Before experiment;Post test:10 weeks end
  The PE entrance examination for senior high school test performance is according to the Sichuan Provincial Department of Education's guidelines for 2022, the scores of high school physical education entrance exams will pass Volleyball dig against the wall; 800m run (Girls); 1000m run (Boys); Pull-ups (girls); Incline pull-ups (girl); Standing Long Jump test. These test taken and quantified on a scale of (10；15；20；25；30；35；40；45；50；55；60；65；70；75；80；85；90；95；100 points). after the test. After the 10-week intervention period, the Investigator will be tested against the assessment metrics, and the Participant's score will be converted to a score that meets this criteria based on the Participant's test results. Each of these tests will be scored according to a standardized scale ranging from 10 to 100 points, with higher scores indicating superior performance.

CONTACTS AND LOCATIONS:
Overall Officials: Yimou MAO, Principal Investigator — Universiti Putra Malaysia
Locations (1):
- Yimou MAO, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No
No Since this is my doctoral thesis experiment, I won't share it until I graduate.

REFERENCES:
- [Background] Pereira A, Costa AM, Santos P, Figueiredo T, Joao PV. Training strategy of explosive strength in young female volleyball players. Medicina (Kaunas). 2015;51(2):126-31. doi: 10.1016/j.medici.2015.03.004. Epub 2015 Apr 1. PMID 25975882
- [Background] Stojanovic D, Momcilovic V, Zadraznik M, Ilic I, Konicanin A, Padulo J, Russo L, Stojanovic T. School-Based TGfU Volleyball Intervention Improves Physical Fitness and Body Composition in Primary School Students: A Cluster-Randomized Trial. Healthcare (Basel). 2023 May 30;11(11):1600. doi: 10.3390/healthcare11111600. PMID 37297741
- [Background] Hu WN, Li DY, Lam WK, Wang Y, Wong DW, Cheung JC. Physical Fitness of Chinese Primary School Students across the Coronavirus (COVID-19) Outbreak: A Retrospective Repeated Cross-Sectional Study. Int J Environ Res Public Health. 2022 Jun 27;19(13):7870. doi: 10.3390/ijerph19137870. PMID 35805528
- See also: This article is from National Library of Medicine. — https://pubmed.ncbi.nlm.nih.gov/25975882/
- See also: This article is from National Library of Medicine. — https://pubmed.ncbi.nlm.nih.gov/37297741/
- See also: This article is from National Library of Medicine. — https://pubmed.ncbi.nlm.nih.gov/35805528/